CLINICAL TRIAL: NCT04944797
Title: Prevalence, Risk Factors and Impact of Anal Incontinence in Patients Followed for Crohn's Disease
Brief Title: Crohn and Anal Incontinence
Acronym: CRIA
Status: Withdrawn | Type: Observational
Why Stopped: The project was abandoned.
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Collaborators: Hôpital Louis Mourier (Other)
Responsible Party: Sponsor
Other Study IDs: CRIA
Record Dates: First submitted 2021-06-15; First posted 2021-06-30 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Anal incontinence affects nearly 5% of the adult population in France. It is defined as the inability for a subject to retain matter and/or gas, outside of voluntary defecation episodes. It results in an uncontrolled loss of gas or stool through the anus. To quantify, anal incontinence clinical scores have been developed of which the most used is the Cleveland score (Jorge and Wexner). A Cleveland score ≥ 5 corresponds to anal incontinence.

Crohn's disease is a chronic inflammatory disease that can affect the entire digestive tract as well as the anus. It leads to destruction of the intestinal wall if not treated early.

The presence of ano-perineal involvement is a factor of severity and poor prognosis of Crohn's disease. The management of these ano-perineal lesions is particularly difficult because of the risks of destruction of the anal sphincter and recurrence of these lesions, as well as the consequences that they induce on anal continence, sexuality and quality of life.

The prevalence of anal incontinence in Crohn's disease has been assessed in three studies by self-questionnaires. In 2013, it was studied in a cohort of British patients followed for chronic inflammatory bowel disease (IBD) (Hemorrhagic rectocolitis or Crohn's disease). Of the 3264 patients who responded to this questionnaire (32.5% of the cohort), 74% claimed to have anal incontinence and in 40% of cases it occurred regularly or a few times. In a study of 184 patients treated at an IBD expert center in Sri Lanka, anal incontinence was reported to be 26%. Only 5 patients reported regular anal incontinence. Vollebregt et al specifically studied the prevalence of anal incontinence in patients followed for Crohn's disease in a Dutch expert center. Of the 325 responses (62%), 20% of patients reported having had an episode of anal incontinence in the last 4 weeks.

In these studies, the prevalence of anal incontinence varies according to the definition of anal incontinence (qualitative or quantitative estimate) and the population studied. No French study has been published on the prevalence of anal incontinence in Crohn's disease.

DETAILED DESCRIPTION:
Many risk factors for anal incontinence have been identified in the general population. In IBD, the risk factors associated with anal incontinence are gender, age, a history of anal stenosis, a history of anal fistula surgery, and a history of colorectal surgery. There is currently only one study that has identified risk factors for anal incontinence specific to Crohn's disease. In this study, the risk factors for anal incontinence were loose stools, a history of colonic or bowel resection related to Crohn's disease, a stenosing phenotype of Crohn's disease, and ano-perineal involvement in Crohn's disease.

The impact of anal incontinence on quality of life is major. Numerous trials show that this handicap is underestimated because of its shameful, embarrassing and intimate nature. The deterioration of quality of life, evaluated by the Inflammatory Bowel Disease Questionnaire (IBDQ) or Fecal Incontinence Quality-of-Life (FIQL) scores, is associated with the severity of anal incontinence in IBD. It is significantly degraded when there are several.

episodes of weekly anal incontinence in patients followed for Crohn's disease. Only one study compared the quality of life of patients with ano-perineal involvement related to Crohn's disease with that of patients with only colonic or intestinal involvement. A significant deterioration in quality of life was reported in those with anoperineal involvement related to Crohn's disease.

One of the therapeutic targets to be achieved in Crohn's disease is the "patient related outcomes" (PRO), i.e. the functional handicap secondary to the disease that is reported by the patient. Anal incontinence is one of the disabilities related to Crohn's disease. The aim of treatment is to stop the handicap and thus to improve the quality of life.

The aim of this study is to evaluate the prevalence, risk factors and impact on quality of life of anal incontinence in a French cohort of patients with Crohn's disease.

ELIGIBILITY:
Inclusion Criteria:

* Patient whose age ≥ 18 years
* French-speaking patient
* Patient followed for Crohn's disease in one of the participating centers (gastroenterology or proctology departments of the Paris-Saint Joseph Hospital Group, gastroenterology department of the Louis Mourier Hospital). The diagnosis of Crohn's disease is based on clinical, endoscopic, radiological and histological criteria.

Exclusion Criteria:

* Patient with a functional stoma
* Patient who objects to participation in the study
* Patient under guardianship or curatorship
* Patient deprived of liberty
* Patient under court protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be offered to consecutively selected patients who meet the eligibility criteria. These patients will be seen in one of the two study centers (gastroenterology and proctology departments at GHPSJ or gastroenterology department at Louis Mourier Hospital):
  * either in day hospital to carry out their treatment (infliximab, adalimumab, vedolizumab, ustekinumab, intravenous iron)
  * or in consultation for their classic follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-03-30 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Determine the prevalence of anal incontinence in patients with Crohn's disease at expert gastroenterology and proctology centers in France. Anal incontinence is defined by a Cleveland or Jorge and Wexner score ≥ 5 | Day 1
  Percentage of patients with Crohn's disease with a Cleveland or Jorge and Wexner score ≥ 5

SECONDARY OUTCOMES:
Compare the prevalence of anal incontinence in patients followed for Crohn's disease on gastroenterology services versus patients followed for ano-perineal involvement in Crohn's disease on a proctology service. | Day 1
  Percentages of patients followed for Crohn's disease in gastroenterology departments (Paris Saint-Joseph Hospital Group and Louis Mourier Hospital) with a Jorge and Wexner score ≥ 5 versus patients followed for ano-perineal involvement of Crohn's disease in a proctology department (Paris Saint-Joseph Hospital Group) with a Jorge and Wexner score ≥ 5
Determine independent risk factors for anal incontinence in Crohn's disease regardless of Crohn's disease location | Day 1
  Analysis of risk factors for anal incontinence
Compare the quality of life of patients with anal incontinence vs. patients without anal incontinence with Crohn's disease | Day 1
  Difference in medians of FIQL quality of life score in patients with anal incontinence vs. patients without anal incontinence with Crohn's disease
Compare the quality of life of patients followed for Crohn's disease on gastroenterology services with anal incontinence versus patients followed for ano-perineal involvement of Crohn's disease on a proctology service with anal incontinence | Day 1
  Difference between the medians of the FIQL quality of life score in patients followed up for Crohn's disease in gastroenterology departments (Groupe hospitalier Paris Saint-Joseph and Hôpital Louis Mourier) and presenting anal incontinence compared to patients followed up for ano-perineal involvement of Crohn's disease in a proctology department (Groupe hospitalier Paris Saint-Joseph) and presenting anal incontinence
Compare the quality of life of patients with anoperineal involvement in Crohn's disease and anal incontinence versus patients with exclusive luminal involvement in Crohn's disease and anal incontinence | Day 1
  Difference in medians of FIQL quality of life score in patients with anoperineal involvement of Crohn's disease and anal incontinence vs. patients with exclusive luminal involvement of Crohn's disease and anal incontinence

CONTACTS AND LOCATIONS:
Overall Officials: Vincent de Parades, MD, Principal Investigator — Fondation Hôpital Saint-Joseph